CLINICAL TRIAL: NCT03858868
Title: Linking Churches With Parks to Increase Physical Activity Among Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: California State University, Los Angeles (Other); San Diego State University (Other)
Responsible Party: Principal Investigator, Kathryn Derose, Senior Policy Researcher, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA218188 (NIH)
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Physical Activity
Keywords: physical activity; community-based health promotion; built environment; faith-based organizations
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Church and park-based intervention (Experimental): Participants at intervention churches will be offered: texting intervention (messages about physical activity); peer leader training; walking groups; park-based fitness classes; sermons; participation in park advisory board; community advocacy.
  Interventions: Behavioral: Church and park-based intervention
- Publicly available physical activity materials (Other): Participants at control churches will be offered standard health educational materials (brochures, tip sheets, posters) about physical activity.
  Interventions: Behavioral: Standard health education on physical activity

INTERVENTIONS:
Behavioral: Church and park-based intervention — Multiple components involving motivational messages and concrete opportunities for physical activity at the church and the local park.
  Arms: Church and park-based intervention
Behavioral: Standard health education on physical activity — Participants will receive publicly available brochures, tip sheets, etc. about physical activity
  Arms: Publicly available physical activity materials

SUMMARY:
This study is a cluster randomized controlled trial of a multi-level intervention that links Latino Catholic churches (n=14) with their local parks to increase physical activity among Latino parishioners (n=1204) in Los Angeles. The study will examine the impact of the intervention on Latino parishioners' PA and health-related outcomes; explore differences in the intervention's effectiveness by gender; and evaluate factors associated with implementation for future dissemination. If successful, the intervention has the potential for sustainability and scale-up across the largest diocese in the U.S. and potentially across the nation.

DETAILED DESCRIPTION:
Engaging in regular physical activity (PA) contributes to positive health outcomes, including longevity, better quality of life, and reduced incidence of cardiovascular diseases, diabetes, depression, certain cancers, and obesity; however, only a minority of U.S. adults meet the minimum guidelines for moderate to vigorous PA (MVPA), and Latinos are less likely than whites to report meeting the guidelines. Public parks comprise local infrastructure that can be leveraged for community PA, but tend to be underutilized, particularly in low-income communities. Parks in low-income and minority communities tend to have less PA programming, especially targeting adults, and higher crime and other factors that affect park use. There is a need for interventions that address community concerns, target the built environment, and "activate" park use. Churches are credible, stable entities that have significant reach within Latino communities and a history of social service provision and advocacy related to health and well-being. The investigators' prior research has found that church-based interventions can be effective across a wide range of health issues and types of churches. This study combines approaches from the research team's extensive prior work with churches and parks to conduct a cluster randomized controlled trial of a multi-level intervention that links Latino Catholic churches (n=14) with their local parks to increase PA among Latino parishioners (n=1204) in Los Angeles. The specific aims are to: (1) Examine the impact of a multi-level church-based intervention that links Catholic parishes to their local parks on Latino parishioners' PA and health-related outcomes (effects on parishioners' MVPA and self-reported PA, heart rate/fitness, waist circumference, waist to hip ratio, body fat, mental health, and perceived social support for PA); (2) Explore differences in the effectiveness of the intervention by gender; and (3) Evaluate factors associated with intervention implementation (facilitators, barriers, fidelity, and replication costs) for future dissemination. The approach targets multiple levels to promote health-enhancing PA through park-based fitness classes led by kinesiology students, peer leader-led walking groups, park-based church events, and church-based PA support activities. It integrates churches' vast social networks, moral authority, and influence with parks' structural and organizational capacity and kinesiology student interns' professional expertise. The intervention makes use of innovative partnerships within and across sectors - faith-based, local parks/city government, and local universities. The inter-sectoral, collaborative approach makes the intervention scalable and sustainable in real-world settings and incorporates action at multiple levels (individuals, churches, and neighborhoods). To the investigators' knowledge, this will be the first study to examine the effectiveness of an integrated church and park-based intervention on Latinos' PA, and it will provide a sustainable model of PA programming in low-income communities. If the intervention proves effective, the increased community capacity through this partnership will lay the groundwork for scale-up across the largest diocese in the U.S. and, potentially, the nation.

ELIGIBILITY:
Inclusion Criteria:

* Does not currently meet physical activity guidelines (150 minutes per week)
* Regularly attends study church
* Does not have health condition that would preclude physical activity

Exclusion Criteria:

* Regularly engages in 150 minutes or more of moderate to vigorous physical activity
* Does not regularly attend study church
* Has health condition that would preclude physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 925 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured physical activity | Change in physical activity between baseline and 12 months
  Accelerometer-assessed moderate to vigorous physical activity at 12 months as compared to baseline

SECONDARY OUTCOMES:
Change in fitness level | Change in fitness level between baseline and 12 months
  Heart rate / fitness as measured by the 3 minute submaximal step test
Change in waist circumference | Change in waist circumference between baseline and 12 months
  Objectively measured waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn P Derose, PhD, MPH, Principal Investigator — RAND
Locations (1):
- RAND Corporation, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported and biometric variables at baseline, 6m and 12m. These will be made available in the form of an electronic database for researchers who successfully complete a registration process. Data will be de-identified and will not contain any direct or indirect identifiers. We will provide a codebook and users must agree to the conditions of use, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Users must submit brief proposals regarding intended use of the data; the study team will determine the scientific soundness of the proposal, as well as whether adequate data protections in place, as part of the decision for the researcher to be able to access the public use dataset.
Time Frame: 6 months after completion of final manuscripts.

REFERENCES:
- [Derived] Derose KP, Cohen DA, Han B, Arredondo EM, Perez LG, Larson A, Loy S, Mata MA, Castro G, De Guttry R, Rodriguez C, Seelam R, Whitley MD, Perez S. Linking churches and parks to promote physical activity among Latinos: Rationale and design of the Parishes & Parks cluster randomized trial. Contemp Clin Trials. 2022 Dec;123:106954. doi: 10.1016/j.cct.2022.106954. Epub 2022 Oct 4. PMID 36206951